CLINICAL TRIAL: NCT01010737
Title: A Phase I/II, Randomized, Single-Blind, Placebo-Controlled Escalating Double-Dose, Safety and Priming Potential Study of an Intramuscular Influenza Vaccine (Multimeric-001) Injected to Elderly Volunteers
Brief Title: A Double-Dose Safety Study of An Influenza Vaccine (Multimeric-001) Injected to Elderly Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BiondVax Pharmaceuticals ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BVX-003
Record Dates: First submitted 2009-10-18; First posted 2009-11-10 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Influenza
Keywords: Multimeric; Vaccine; Influenza; elderly; phase 1/2; safety; efficacy; tolerability; reactogenicity; Montanide; hemagglutinin inhibition; HAI; TIV
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Multimeric-001 250 mcg (Experimental): 250mcg of Multimeric-001 was administered twice at an interval of 19-23 days via the IM route to 10 participants as a primer and then a TIV boost was administered.
  Interventions: Biological: Multimeric-001 250 mcg; Biological: TIV
- Adjuvant: Montonide isa 51 VG (Active Comparator): Adjuvanted PBS was administered twice with a 19-23 day interval via the IM route to 10 participants and then a TIV boost was administered.
  Interventions: Biological: Adjuvant: Montonide isa 51 VG; Biological: TIV
- Placebo (Active Comparator): PBS was administered twice with a 19-23 day interval via the IM route to 10 participants and then a TIV boost was administered.
  Interventions: Biological: Adjuvant: Montonide isa 51 VG; Biological: TIV
- Multimeric-001 500 mcg (Experimental): 500mcg of M-001 was administered twice with an interval of 19-23 days via the IM route to 10 participants as a primer and then a TIV boost was administered.
  Interventions: Biological: Adjuvanted Multimeric-001 500mcg; Biological: TIV
- Adjuvanted Multimeric-001 500mcg (Experimental): 5000mcg of Adjuvanted M-001 was administered twice with an interval of 19-23 days via the IM route to 10 participants as a primer and then a TIV boost was administered.
  Interventions: Biological: Adjuvanted Multimeric-001 250mcg; Biological: TIV
- Adjuvanted Multimeric-001 250mcg (Experimental): 250mcg of Adjuvanted M-001 was administered twice with an interval of 19-23 days via the IM route to 10 participants as a primer and then a TIV boost was administered.
  Interventions: Biological: Placebo; Biological: Multimeric-001 500 mcg; Biological: TIV

INTERVENTIONS:
Biological: Multimeric-001 250 mcg — Multimeric-001 (M-001) was administered twice at a dose of 250mcg via the IM route to 10 participants as a primer, followed by TIV boost immunization. in 19-23 days interval between them.
  Arms: Multimeric-001 250 mcg
Biological: Adjuvanted Multimeric-001 250mcg — Injection of Multimeric-001 250 mcg with Adjuvant Montonide isa 51 VG, 2 doses with interval of 19-23 days between them
  Arms: Adjuvanted Multimeric-001 500mcg
Biological: Placebo — Placebo injected with PBS (Phosphate Buffered Saline), 2 injections with the interval of 19-23 days between them.
  Arms: Adjuvanted Multimeric-001 250mcg
Biological: Adjuvant: Montonide isa 51 VG — Injection of Placebo with Adjuvant Montonide isa 51 VG, 2 injections with the interval of 19-23 days between them.
  Arms: Adjuvant: Montonide isa 51 VG; Placebo
Biological: Multimeric-001 500 mcg — Injection of Multimeric-001 with PBS, 2 injections with the interval of 19-23 days between them.
  Arms: Adjuvanted Multimeric-001 250mcg
Biological: Adjuvanted Multimeric-001 500mcg — Injection of Multimeric-001 500 mcg with Adjuvant Montonide isa 51 VG, 2 doses with the interval of 19-23 days between them
  Arms: Multimeric-001 500 mcg
Biological: TIV — Injection of the conventional flu vaccine: Vaxigrip to all study participants.
  Other Names: Vaxigrip

SUMMARY:
This is a phase I/II, randomized, single-blind, placebo-controlled escalating double-dose study of the safety and priming potential of an intramuscular Influenza vaccine (Multimeric-001) injected to elderly volunteers.

DETAILED DESCRIPTION:
This is a Phase I/II single-center, randomized, placebo-controlled, single-blind, dose-escalation, double-dose administration study comprising two dosing cohorts (Cohort 1: 250 mcg M-001 per injection and Cohort 2: 500 mcg M-001 per injection) with 20 subjects in each cohort receiving either adjuvanted or non-adjuvanted formulations. The adjuvant used was Montanide ISA VG51. Cohort 3 with 20 subjects was administered placebo. After priming with M-001 or placebo, all participants were administered a boost of a conventional trivalent vaccine on day 42.

There was a minimum of 10 days interval between last dosing of the first injection to the last subject of the 250 μg cohort (Cohort 1) and first dosing of the first subject injection with 500 µg cohort (Cohort 2).

For each subject, the second injection was performed 21+2 days after his/her first injection, provided they were deemed fit to be dosed by a study physician.

The DSMB reviewed the safety data obtained from cohorts 1 and 2 before approving their second injection and before dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the age of 55 and 75 years (inclusive):

  * Healthy or treated for any or all of the following conditions:

    * Hypertension, under control with standard medications
    * Hyperlipidemia, medically treated
* Subjects who provide written informed consent to participate in the study.
* Subjects able to adhere to the visit schedule and protocol requirements and be available to complete the study.
* Haematology, chemistry and urinalysis values with no clinical significance or do not reflect a medical condition which, according to the physician's judgment, might confound the results of the study or pose additional risk to the subject by participation in the study.
* Female of childbearing age must agree to use an acceptable method of contraception and male subjects should use a condom throughout the study period (including the follow up- where applicable) if female partner is not using an effective contraceptive method.

Exclusion Criteria:

* Known history of significant medical disorder, which in the investigator's judgment, might confound the results of the study or pose additional risk to the subject by participation in the study.
* Renal dysfunction.
* COPD.
* Chronic cardiovascular system disorders (except hypertension adequately controlled by standard medications).
* Asthma
* Diabetes mellitus.
* Subjects with known Guillain Barré Syndrome in the past.
* Two or more hospitalizations within the last year prior to screening visit.
* Bleeding disorders including hemophilia or thrombocytopenia, or treatment with anticoagulant therapy (risk of bleeding with intramuscular injection).
* Immunocompromised patients and those receiving concomitant immunosuppressive therapy; or other immune modulating drugs including chronic steroid treatment.
* Subjects who have been immunized with anti-influenza vaccine or infected by influenza virus within eight months prior to the screening visit.
* Administration of any vaccine 30 days before the screening visit.
* Known hypersensitivity to previous influenza vaccination.
* Use of an influenza antiviral medication within 4 weeks of vaccination.
* Known hypersensitivity and/or allergy to any drug or vaccine.
* Known hypersensitivity to egg proteins (eggs or egg products), chicken proteins, or any of the vaccine components, in particular, neomycin, formaldehyde, and octoxinol 9,
* Known history of drug or alcohol abuse.
* Any clinically significant abnormality upon physical examination or in the clinical laboratory tests at screening visit which, according to the physician's judgment, might confound the results of the study or pose additional risk to the subject by participation in the study.
* Increased liver enzymes more than 2.5 times above the upper reference level.
* Positive serology for HIV, HCV antibody or HBsAg.
* Any acute medical situation (e.g. acute infection, ongoing flu symptoms) with or without fever within 48 hours of vaccination, which is considered of significance by the Principal Investigator.
* Pregnant or lactating women at entry to study and those who are unwilling to agree to continue to use acceptable methods of contraception for two months after completion of the study (if applicable).
* Positive blood pregnancy test on screening.
* Subjects who participated in another clinical study within 30 days prior to study entry.
* Subjects who are non-cooperative or unwilling to sign consent form.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety, local and systemic tolerability and reactogenicity of Multimeric-001 vaccine when administered intramuscularly twice to elderly male and female subjects, using chemistry, CBC, fibrinogen, and urinalysis measurements. | From day 0 until termination visit
  The Multimeric-001 vaccine exhibits a positive safety profile. The number of subjects reporting adverse events (AEs) after treatment with active vaccines was similar to respective placebo cohorts. Overall AE frequencies for each active group were similar to those of placebo counterparts.

SECONDARY OUTCOMES:
To characterize the immune response | 21 days after second immunization with M-001 and 21 days after TIV boost
  The Multimeric-001 vaccine induces both humoral and cellular immune responses, confirming previous findings in younger adults.
To monitor cellular immune responses | 21 days after second M-001 immunization
  PBMC proliferation associated with IFN gamma secretion was detected after prime immunizations following in vitro exposure of the cells to M-001 or influenza viruses.
To obtain preliminary data on the contribution of the adjuvant | 21 days after second M-001 immunization and 21 days after TIV boost
  Adjuvant had an impact on anti-M-001 IgG levels but not on HAI antibody levels.
To obtain preliminary evidence about the efficacy of M-001 as a primer | 21 days after TIV boost
  The prime-boost regimen elicits HAI immune responses, which enables assessment of an accepted surrogate marker considered to correlate with influenza vaccine activity.Priming with M-001 before a TIV boost resulted in a greater proportion of subjects seroconverted to TIV and non-TIV strains as compared to subjects given TIV alone.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, MD, Principal Investigator — CRC, Sourascky MC, Israel
Locations (1):
- Tasmc Crc, Tel Aviv, Israel